CLINICAL TRIAL: NCT07250022
Title: Detection of Residual Caries on Class II Cavity Walls in Primary Teeth Following Atraumatic Restorative Treatment (ART): A Comparative Evaluation of Fluorescence-Aided Caries Excavation (FACE), Caries Detection Dye, and Clinical Assessment
Brief Title: Detection of Residual Caries on Class II Cavity Walls in Primary Teeth Following Atraumatic Restorative Treatment (ART)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Burak Carıkcıoglu, Associate Professor, Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: COMU-BCARIKCIOGLU-2025
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Primary Dental Caries
Keywords: dentin caries; dental atraumatic restorative treatment; primary teeth; FACE; residual caries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FACE + Caries Detection Dye (Active Comparator)
  Interventions: Diagnostic Test: FACE + Caries Detection Dye
- FACE + Visual-Tactile Examination (Active Comparator)
  Interventions: Diagnostic Test: FACE + Visual-Tactile Examination

INTERVENTIONS:
Diagnostic Test: FACE + Caries Detection Dye — Residual caries detection performed using FACE and caries detection dye.
  Arms: FACE + Caries Detection Dye
Diagnostic Test: FACE + Visual-Tactile Examination — Residual caries detection performed using FACE and visual-tactile method.
  Arms: FACE + Visual-Tactile Examination

SUMMARY:
The primary aim of this study is to compare the diagnostic agreement and effectiveness of three different methods-Fluorescence-Aided Caries Excavation (FACE), caries detection dye, and clinical observation-in detecting residual caries remaining on cavity walls of primary teeth following Atraumatic Restorative Treatment (ART). Through this comparison, the study seeks to identify the method that provides more reliable and accurate results, thereby contributing to clinical practice by guiding clinicians and supporting the development of strategies to enhance the long-term success of ART.

DETAILED DESCRIPTION:
Effective management of dental caries in primary teeth is of great importance for pain relief, infection prevention, and the maintenance of a child's overall health. Atraumatic Restorative Treatment (ART), which is frequently preferred in pediatric patients and in regions with limited resources, is a minimally invasive approach that involves the selective removal of carious tissue using hand instruments instead of rotary tools, followed by restoration of the cavity with glass ionomer cement. This method aims to preserve tooth structure, enhance patient comfort, and reduce pulpal irritation. However, the primary limitation of ART is that caries removal relies on the clinician's visual and tactile assessment. This subjectivity increases the risk of residual caries remaining on the cavity walls, which can negatively affect the success and long-term durability of the restoration. The presence of a larger pulp chamber and thinner dentin structure in primary teeth further exacerbates this risk.

Reliable detection of residual caries is therefore crucial to the success of ART. Nevertheless, traditional methods such as clinical observation and caries detection dyes have notable limitations. Clinical observation is subject to low reproducibility due to its dependence on individual experience and judgment, while caries detection dyes can stain not only infected dentin but also demineralized yet healthy tissue, potentially leading to unnecessary tissue removal and an increased risk of pulp exposure. This outcome contradicts the minimally invasive philosophy of ART. Consequently, the use of more objective and precise techniques, such as Fluorescence-Aided Caries Excavation (FACE), has gained increasing importance for accurate detection of residual caries and improvement of treatment outcomes.

Participants in this study will consist of children aged 4 to 9 years who are medically healthy and capable of cooperating during the examination. Each primary molar will be evaluated in six distinct regions: axial wall, gingival floor, enamel-dentin junction, buccal wall, lingual wall, and pulpal wall. The assessment will be conducted sequentially using three different methods: Fluorescence-Aided Caries Excavation (FACE), caries detection dye (Caries Detector, Kuraray, Okayama, Japan), and clinical observation. The FACE method will be performed in a non-contact manner using the D-light Pro GC device (DT mode, GC Europe NV, Leuven, Belgium). The other two methods will involve visual-tactile examination under standard clinical conditions.

All evaluations will be carried out under identical conditions by two independent observers, and each cavity wall will be recorded as either "caries present" or "caries absent." The collected data will be transferred to the SPSS software for statistical analysis and coded as 1/0 (present/absent). In addition, participants' age, gender, dmft index, tooth location (maxilla/mandible), and tooth type (first or second primary molar) will be documented. These variables will allow for the statistical evaluation of potential demographic and clinical factors associated with the presence of residual caries. After the application of all three diagnostic methods on the same cavity, if any of the techniques indicated the presence of residual caries, the clinician-at their discretion-performed additional excavation to remove the affected tissue before proceeding to the final restoration. All teeth were subsequently restored using high-viscosity glass ionomer cement, in accordance with the ART protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age 4-9 years at enrollment
* Healthy children who can cooperate with dental examination
* Multi-surface carious cavities that are asymptomatic (no acute symptoms)
* Written informed consent from parent/guardian and assent from the child

Exclusion Criteria:

* Acute dental infection present
* Any systemic disease/condition
* Lack of cooperation during the procedure
* Refusal to participate / informed consent not obtained from parent/guardian and/or assent not obtained from the child

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 212 (Estimated)
Dates: Start 2025-12-20 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of residual caries detection accuracy using FACE and caries detector dye versus FACE and visual-tactile examination | Baseline (immediately after caries removal procedure; single visit; up to 10 minutes; no follow-up required)
  Residual caries detection will be performed in two diagnostic arms: (1) FACE combined with caries detector dye and (2) FACE combined with visual-tactile examination. After atraumatic caries removal, the presence or absence of residual caries will be evaluated on six cavity walls (axial, gingival, enamel-dentin junction, buccal, lingual, and pulpal). Diagnostic accuracy will be expressed as sensitivity, specificity, and overall accuracy compared with a reference standard (soft dentin confirmed by tactile evaluation).

SECONDARY OUTCOMES:
Assessment of residual caries detection by visual-tactile examination | Baseline (immediately after caries removal procedure; up to 5 minutes; no follow-up required)
  Visual-tactile inspection will assess color, hardness, and texture of the dentin surface. Soft or dark dentin areas, or those producing a "catch" when probed, will be considered positive for residual caries.
Assessment of residual caries detection by caries detector dye | Baseline (immediately after caries removal procedure; up to 10 minutes; no follow-up required)
  Caries detector dye (Caries Detector, Kuraray, Japan) will be applied for 10 seconds and rinsed. Areas showing red or pink staining will be classified as residual caries.
Assessment of residual caries detection by FACE (Fluorescence-Aided Caries Excavation) | Baseline (immediately after caries removal procedure; up to 10 minutes; no follow-up required)
  Using the D-Light Pro device (GC Europe), cavity walls will be examined under violet-blue excitation light. Red-orange fluorescence areas will be identified as residual caries; green fluorescence areas will be considered sound dentin.
Assessment of residual caries detection rate per cavity wall | Baseline (immediately after caries removal procedure; up to 10 minutes; no follow-up required)
  For each cavity, residual caries presence (yes/no) will be recorded in six specific regions (axial, gingival, enamel-dentin junction, buccal, lingual, and pulpal). The percentage of positive areas will be calculated for each diagnostic method.

CONTACTS AND LOCATIONS:
Overall Officials: Burak Çarıkçıoğlu, Associate Professor, Principal Investigator — Çanakkale Onsekiz Mart University; Hilal Öztürk, Research Assistant, Principal Investigator — Çanakkale Onsekiz Mart University; İDİL AY ŞİMŞEK, Research Assistant, Principal Investigator — Çanakkale Onsekiz Mart University
Locations (1):
- Canakkale Onsekiz Mart University, Çanakkale, Kepez, Turkey (Türkiye)